CLINICAL TRIAL: NCT04817865
Title: A Retrospective Comparison of Pre-procedural PCR and Culture-based UTI Assessment Prior to Intravesical Botox for the Treatment of Neurogenic or Non-neurogenic Overactive Bladder
Brief Title: Comparison of Pre-procedural PCR and Culture-based UTI Assessment Prior to Intravesical Botox Injection
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor's decision
Sponsor: Pathnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-btxuti
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Urinary Tract Infections
Keywords: Overactive Bladder; PCR; Urine Culture; Botox Injection
MeSH Terms: conditions — Urinary Tract Infections; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Pre-Procedural Urine Culture: This is a control cohort that follows standard pre-procedural protocol by implementing antibiotic prophylaxis and treatment regimens based on dipstick urine analysis (UA) followed by reflexed traditional urine culture and sensitivity (C&S) methods performed before injection.
  Interventions: Diagnostic Test: Urine Culture
- Pre-Procedural M-PCR/P-AST: This is an experimental cohort that implements Multiplex-PCR with Pooled Antibiotic Susceptibility Testing (M-PCR/P-AST) for pre-procedural UTI screening. The cohort follows an antibiotic treatment regimen based on the results of M-PCR/P-AST.
  Interventions: Diagnostic Test: Multiplex-PCR with Pooled Antibiotic Susceptibility Testing (M-PCR/P-AST)

INTERVENTIONS:
Diagnostic Test: Multiplex-PCR with Pooled Antibiotic Susceptibility Testing (M-PCR/P-AST) — M-PCR/P-AST is a dual assessment test that detects pathogenic DNA commonly associated with urinary tract infections and identifies their genotypic and phenotypic antibiotic resistance.
  Groups: Pre-Procedural M-PCR/P-AST
Diagnostic Test: Urine Culture — A traditional clinical UTI evaluation consisting of non-molecular standard urine culture (SUC) and sensitivity testing methods.
  Groups: Standard Pre-Procedural Urine Culture

SUMMARY:
This study is a retrospective record review to determine whether a novel multiplex PCR assay can be utilized as a screening method for UTI in patients receiving Botox injection to treat overactive bladder (OAB).

DETAILED DESCRIPTION:
The novel multiplex real-time PCR assay with mixed floral antibiotic resistance profiling offers a higher degree of sensitivity and specificity than conventional culture methods in the identification of UTI pathogens as determined by a previous prospective comparison study. This is a retrospective record review comparing PCR and culture-based assessments for UTI in patients receiving Botox injection to treat overactive bladder (OAB). Investigators aim to determine whether M-PCR/P-AST can be utilized as a screening method for UTI in these patients and whether whether antibiotic prophylaxis, peri-procedural antibiotics, and post-injection antibiotic therapy based on patients' pre-procedural M-PCR/P-AST results in improved response to Botox injection compared to standard of care. The attributes and advantages of PCR testing over the use of traditional urine cultures, and the potential identification of polymicrobial infections with complicated resistance sharing mechanisms, may significantly improve patient care.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Subject is male or female
* >18 years of age at date of injection
* Subject receiving BoNT injection for symptoms of OAB (including urgency, urinary incontinence, and detrusor overactivity) refractory to first-line therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving Botox injections for the treatment of neurogenic or non-neurogenic OAB
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Post procedural UTI | Up to 3 weeks post injection
  Defined as development of UTI confirmed by urine culture/PCR in the setting of UTI symptoms requiring antibiotic therapy
Recurrent UTI | Up to 12 months post-injection
  Defined as the development of multiple UTI confirmed by urine culture/PCR in the setting of UTI symptoms requiring antibiotic therapy
Resistant UTI | Up to 12 months post-injection
  Defined as UTI that manifests as a persistence or worsening of symptoms during antibiotic course
Antibiotic Usage | Up to 3 weeks post-injection
  Defined as total number of post-procedural antibiotics ordered/taken within 3 weeks post BOTOX injection
Visit Reschedule/Cancellation Rate | Up to 1 year after pre-procedural assessment
  Defined as any injection visit cancelled/postponed/rescheduled due to results of preprocedural assessments (abnormal UA, lower urinary tract symptoms etc.)

SECONDARY OUTCOMES:
UTI-related ED Visit Rate | Up to 3 weeks post-injection
  Defined as any visit to the ED relating to symptoms of UTI within 3 weeks post-Botox injection
UTI-hospital Admission Rate | Up to 3 weeks post-injection
  Defined as any admission to the hospital (from home/ED or clinic transfer) relating to symptoms of UTI within 3 weeks post-Botox injection

CONTACTS AND LOCATIONS:
Overall Officials: David Baunoch, PhD, Principal Investigator — Pathnostics, Inc.
Locations (1):
- Comprehensive Urologic Care, Barrington, Illinois, United States

IPD SHARING:
Plan to Share IPD: No